CLINICAL TRIAL: NCT04283188
Title: Pragmatic Patient-Oriented 12-Month Extension Study of Dialectical Behavior Therapy for Youth With Bipolar Disorder
Brief Title: 12-Month Extension Study of Dialectical Behavior Therapy for Youth With Bipolar Disorder
Acronym: DB2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: University of Pittsburgh (Other); Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Dr. Benjamin Goldstein, Director of the Centre for Youth Bipolar Disorder, Senior Scientist, Psychiatrist, Principal Investigator, Professor of Psychiatry, Pharmacology & Toxicology, and Psychological Clinical Science, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 447-2019; 151/2020 (Other: Centre for Addiction and Mental Health Research Ethics Board)
Record Dates: First submitted 2020-02-19; First posted 2020-02-25 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Bipolar Disorder
Keywords: Dialectical behavior therapy
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adolescents with bipolar disorder (Experimental): 25 adolescents aged 14 to 21 with bipolar disorder (type I, type II, not otherwise specified/nos) will be enrolled in the dialectical behavioral therapy intervention.
  Interventions: Behavioral: Dialectical behavioral therapy

INTERVENTIONS:
Behavioral: Dialectical behavioral therapy — Participants will be provided with the option to continue treatment with their study therapist. For those who elect to continue with DBT sessions, they will discuss frequency of sessions with their therapist, in addition to selecting type of sessions (individual and/or family skills). Participants who elect not to continue with DBT sessions at the time of enrollment will retain the option of being able to request additional sessions at any point during the 12-month study. Irrespective of participation in additional DBT sessions, all participants will be asked to complete follow-up interviews and questionnaires.
  Other Names: DBT

SUMMARY:
The overarching goal of this project is to evaluate the longer-term effects of implementing DBT for adolescents with BD in a subspecialty clinic. In collaboration with the University of Pittsburgh and continuing from the parent study (042-2018), this study will measure the longer-term effects of DBT in additional the the longer-term effects of DBT training on study therapist knowledge and performance.

DETAILED DESCRIPTION:
This is an extension study related to an ongoing implementation study of dialectical behavior therapy (DBT) for adolescents with bipolar disorder, in collaboration with investigators at the University of Pittsburgh. During the conduct of that initial study (the DITO study; REB PIN 042-2018), compelling questions have been raised by the investigators, study therapists, and participants/patients about what will happen following participation in the initial study: Which DBT outcomes are sustained over time? Will patients request and/or require additional booster sessions? Will study therapists remain adherent to the treatment model? There is sparse knowledge regarding what happens after a course of DBT is completed, and this study seeks to advance our understanding of what happens in the year after DBT by addressing these questions. This study provides a unique opportunity to examine the frequency, dose, and indications for ongoing DBT treatment for participants who have completed one year of DBT at the Centre for Youth Bipolar Disorder (CYBD). In the spirit of the original dissemination and implementation study, this study is focused on "real-world" issues routinely faced by study therapists and patients, and anticipated findings will inform future randomized controlled trials on this topic.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Age 14 years, 0 months to 21 years, 11 months
* Meet diagnostic criteria for BD by KSADS-PL
* Followed by a CAMH or Sunnybrook psychiatrist who provides ongoing care
* If BD-I, taking ≥1 mood stabilizing medication (i.e., antimanic anticonvulsant, antipsychotic, and/or lithium
* Has completed participation in the DITO study (REB PIN 042-2018)
* Able and willing to give informed consent/assent to participate.

Exclusion Criteria:

* Evidence of mental retardation, moderate to severe pervasive developmental disorder, or organic central nervous system disorder by the K-SADS-PL, parent report, medical history, or school records
* A life-threatening medical condition requiring immediate treatment
* Current victim of sexual or physical abuse.

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2020-02-19 (Actual); Primary Completion 2022-11-18 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
Therapist satisfaction and acceptability | 18 months
  Therapists will complete a questionnaire (Therapist Satisfaction and Acceptability Questionnaire) assessing their satisfaction with the training and treatment approach at 6 months. Acceptability will be defined as mean acceptability ratings > 5 ("acceptable") on a likert scale from 1 ("very unacceptable") to 7 ("very acceptable").
Therapist satisfaction and acceptability | 24 months
  Therapists will complete a questionnaire (Therapist Satisfaction and Acceptability Questionnaire) assessing their satisfaction with the training and treatment approach at 6 months. Acceptability will be defined as mean acceptability ratings > 5 ("acceptable") on a likert scale from 1 ("very unacceptable") to 7 ("very acceptable").
Therapists will adhere to the Dialectical Behavior Therapy Adherence Rating Scale | Through study completion (three years), an average of semi-annually.
  Tapes will be rated for adherence using the Dialectical Behavior Therapy (DBT) Adherence Rating scale. The scale generates a Global Score of DBT adherence and subscale scores for the 12 DBT strategy domains. To examine sustained adherence, each therapist will submit 3 consecutive sessions for adherence coding. The rating scale is not available to the public and is utilized by the DBT-Linehan Board of Certification (copyright). Please see http://www.dbt-lbc.org/downloads/Applicant_Handbook_final_with_RW_review_2018.pdf for more information.
Change in symptoms using the Longitudinal Interval Follow-up Evaluation (LIFE) | 12 months to 18 months
  The Longitudinal Interval Follow-up Evaluation (LIFE) will provide a comprehensive cross-sectional and longitudinal picture of the symptomatic and psychosocial course and outcome of all participants in this study. Scores range from 0-3 on certain disorders and 0-6 for other disorders. High scores indicate high level of symptom impairment.
Change in symptoms using the Longitudinal Interval Follow-up Evaluation (LIFE) | 18 months to 24 months
  The Longitudinal Interval Follow-up Evaluation (LIFE) will provide a comprehensive cross-sectional and longitudinal picture of the symptomatic and psychosocial course and outcome of all participants in this study. Scores range from 0-3 on certain disorders and 0-6 for other disorders. High scores indicate high level of symptom impairment.
Change in hypo/mania symptoms using the Child Mania Rating Scale (CMRS) | 12 months to 15 months
  Parent and adolescent reported depressive and manic symptoms will be measured via the Child Mania Rating Scale (CMRS). The CMRS is a valid 21-item screening instrument, reflecting the DSM-IV criteria for a manic episode, with each response rated on a four-point Likert-type scale with scores ranging from 0 to 3. High scores indicate higher level of symptoms.
Change in hypo/mania symptoms using the Child Mania Rating Scale (CMRS) | 15 months to 18 months
  Parent and adolescent reported depressive and manic symptoms will be measured via the Child Mania Rating Scale (CMRS). The CMRS is a valid 21-item screening instrument, reflecting the DSM-IV criteria for a manic episode, with each response rated on a four-point Likert-type scale with scores ranging from 0 to 3. High scores indicate higher level of symptoms.
Change in hypo/mania symptoms using the Child Mania Rating Scale (CMRS) | 18 months to 121 months
  Parent and adolescent reported depressive and manic symptoms will be measured via the Child Mania Rating Scale (CMRS). The CMRS is a valid 21-item screening instrument, reflecting the DSM-IV criteria for a manic episode, with each response rated on a four-point Likert-type scale with scores ranging from 0 to 3. High scores indicate higher level of symptoms.
Change in hypo/mania symptoms using the Child Mania Rating Scale (CMRS) | 21 months to 24 months
  Parent and adolescent reported depressive and manic symptoms will be measured via the Child Mania Rating Scale (CMRS). The CMRS is a valid 21-item screening instrument, reflecting the DSM-IV criteria for a manic episode, with each response rated on a four-point Likert-type scale with scores ranging from 0 to 3. High scores indicate higher level of symptoms.
Change in suicidality using the Columbia-Suicide Severity Rating Scale (C-SSRS) | 12 months to 18 months
  We will assess suicidal events (past and over follow-up) with the Pediatric Version of the Columbia-Suicide Severity Rating Scale (C-SSRS). The C-SSRS has sound psychometric properties, yields ratings of widely accepted definitions of youth suicidal events, and was used in other pediatric treatment trials yielding standardized outcomes to compare across studies. This is a semi-structured interview that includes yes/no questions as well as narrative. It captures number of suicidal events as well as type and severity.
Change in suicidality using the Columbia-Suicide Severity Rating Scale (C-SSRS) | 18 months to 24 months
  We will assess suicidal events (past and over follow-up) with the Pediatric Version of the Columbia-Suicide Severity Rating Scale (C-SSRS). The C-SSRS has sound psychometric properties, yields ratings of widely accepted definitions of youth suicidal events, and was used in other pediatric treatment trials yielding standardized outcomes to compare across studies. This is a semi-structured interview that includes yes/no questions as well as narrative. It captures number of suicidal events as well as type and severity.
Change in symptoms using the Mood and Feelings Questionnaire (MFQ) | 12 months to 15 months
  Self-reported depressive and manic symptoms will be measured via the Mood and Feelings Questionnaire (MFQ). Responses are made on a 3-point scale ("0=not true", "1=sometimes true" and "2=true").
Change in symptoms using the Mood and Feelings Questionnaire (MFQ) | 15 months to 18 months
  Self-reported depressive and manic symptoms will be measured via the Mood and Feelings Questionnaire (MFQ). Responses are made on a 3-point scale ("0=not true", "1=sometimes true" and "2=true").
Change in symptoms using the Mood and Feelings Questionnaire (MFQ) | 18 months to 21 months
  Self-reported depressive and manic symptoms will be measured via the Mood and Feelings Questionnaire (MFQ). Responses are made on a 3-point scale ("0=not true", "1=sometimes true" and "2=true").
Change in symptoms using the Mood and Feelings Questionnaire (MFQ) | 21 months to 24 months
  Self-reported depressive and manic symptoms will be measured via the Mood and Feelings Questionnaire (MFQ). Responses are made on a 3-point scale ("0=not true", "1=sometimes true" and "2=true").
Change in suicidality using the Suicidal Ideation Questionnaire (SIQ) | 12 months to 15 months
  Adolescents will also complete the self-report Suicidal Ideation (SIQ), which is intended to identify adolescents whose level of suicidal ideation is severe enough to warrant further intervention. Each item is rated on a 7-point Likert-type scale (0= "I never had this thought" to 6="almost every day") and is used to indicate the frequency with which the adolescent experiences each thought.
Change in suicidality using the Suicidal Ideation Questionnaire (SIQ) | 15 months to 18 months
  Adolescents will also complete the self-report Suicidal Ideation (SIQ), which is intended to identify adolescents whose level of suicidal ideation is severe enough to warrant further intervention. Each item is rated on a 7-point Likert-type scale (0= "I never had this thought" to 6="almost every day") and is used to indicate the frequency with which the adolescent experiences each thought.
Change in suicidality using the Suicidal Ideation Questionnaire (SIQ) | 18 months to 21 months
  Adolescents will also complete the self-report Suicidal Ideation (SIQ), which is intended to identify adolescents whose level of suicidal ideation is severe enough to warrant further intervention. Each item is rated on a 7-point Likert-type scale (0= "I never had this thought" to 6="almost every day") and is used to indicate the frequency with which the adolescent experiences each thought.
Change in suicidality using the Suicidal Ideation Questionnaire (SIQ) | 21 months to 24 months
  Adolescents will also complete the self-report Suicidal Ideation (SIQ), which is intended to identify adolescents whose level of suicidal ideation is severe enough to warrant further intervention. Each item is rated on a 7-point Likert-type scale (0= "I never had this thought" to 6="almost every day") and is used to indicate the frequency with which the adolescent experiences each thought.
Change in emotion regulation using the Difficulties in Emotion Regulation Scale (DERS) | 12 months to 15 months
  Adolescents will also complete the Difficulties in Emotion Regulation (DERS), a 36-item questionnaire assessing emotional dysregulation. Participants indicate how often each item applies to them on a scale from 1="almost never; 0-10 percent" to 5= "almost always; 91-100 percent".
Change in emotion regulation using the Difficulties in Emotion Regulation Scale (DERS) | 15 months to 18 months
  Adolescents will also complete the Difficulties in Emotion Regulation (DERS), a 36-item questionnaire assessing emotional dysregulation. Participants indicate how often each item applies to them on a scale from 1="almost never; 0-10 percent" to 5= "almost always; 91-100 percent".
Change in emotion regulation using the Difficulties in Emotion Regulation Scale (DERS) | 18 months to 21 months
  Adolescents will also complete the Difficulties in Emotion Regulation (DERS), a 36-item questionnaire assessing emotional dysregulation. Participants indicate how often each item applies to them on a scale from 1="almost never; 0-10 percent" to 5= "almost always; 91-100 percent".
Change in emotion regulation using the Difficulties in Emotion Regulation Scale (DERS) | 21 months to 24 months
  Adolescents will also complete the Difficulties in Emotion Regulation (DERS), a 36-item questionnaire assessing emotional dysregulation. Participants indicate how often each item applies to them on a scale from 1="almost never; 0-10 percent" to 5= "almost always; 91-100 percent".
Treatment Satisfaction Questionnaire (18-item) | 15 months
  Following the year-long DBT intervention, patients and parents will complete an 18-item Treatment Satisfaction Questionnaire. This assesses clients' satisfaction of the service (responses range from quite dissatisfied to very satisfied) as well as whether or not the service addressed the clients' needs.
Treatment Satisfaction Questionnaire (18-item) | 18 months
  Following the year-long DBT intervention, patients and parents will complete an 18-item Treatment Satisfaction Questionnaire. This assesses clients' satisfaction of the service (responses range from quite dissatisfied to very satisfied) as well as whether or not the service addressed the clients' needs.
Treatment Satisfaction Questionnaire (18-item) | 21 months
  Following the year-long DBT intervention, patients and parents will complete an 18-item Treatment Satisfaction Questionnaire. This assesses clients' satisfaction of the service (responses range from quite dissatisfied to very satisfied) as well as whether or not the service addressed the clients' needs.
Treatment Satisfaction Questionnaire (18-item) | 24 months
  Following the year-long DBT intervention, patients and parents will complete an 18-item Treatment Satisfaction Questionnaire. This assesses clients' satisfaction of the service (responses range from quite dissatisfied to very satisfied) as well as whether or not the service addressed the clients' needs.
Change in symptoms using the Structured Interview for DSM-IV Personality (SIDP-IV): Borderline Personality Disorder | 12 months to 18 months
  Borderline and antisocial personality symptoms will be assessed using the Structured Interview for DSM-IV Personality. The SID-P uses a semi structured interview format to assess for symptoms of personality disorders. Scores one each item range from 0 to 3 and high scores indicate symptoms of borderline personality disorder and levels of impairment.
Change in symptoms using the Structured Interview for DSM-IV Personality (SIDP-IV): Borderline Personality Disorder | 18 months to 24 months
  Borderline and antisocial personality symptoms will be assessed using the Structured Interview for DSM-IV Personality. The SID-P uses a semi structured interview format to assess for symptoms of personality disorders. Scores one each item range from 0 to 3 and high scores indicate symptoms of borderline personality disorder and levels of impairment.
Change in affective lability using the Children's Affective Lability Scale (CALS) | 12 months to 15 months
  The Children's Affective Lability Scale (CALS) is a reliable 20-item adolescent- and parent-reported measure of mood lability, derived from the adult Affective Lability Scale that was specifically designed for adults with BD. It yields a total score as well as an angry/depressed factor and a disinhibited/impersistent factor.
Change in affective lability using the Children's Affective Lability Scale (CALS) | 15 months to 18 months
  The Children's Affective Lability Scale (CALS) is a reliable 20-item adolescent- and parent-reported measure of mood lability, derived from the adult Affective Lability Scale that was specifically designed for adults with BD. It yields a total score as well as an angry/depressed factor and a disinhibited/impersistent factor. Item scores range from 0 to 4 and higher scores indicate higher affective lability.
Change in affective lability using the Children's Affective Lability Scale (CALS) | 18 months to 21 months
  The Children's Affective Lability Scale (CALS) is a reliable 20-item adolescent- and parent-reported measure of mood lability, derived from the adult Affective Lability Scale that was specifically designed for adults with BD. It yields a total score as well as an angry/depressed factor and a disinhibited/impersistent factor. Item scores range from 0 to 4 and higher scores indicate higher affective lability.
Change in affective lability using the Children's Affective Lability Scale (CALS) | 21 months to 24 months
  The Children's Affective Lability Scale (CALS) is a reliable 20-item adolescent- and parent-reported measure of mood lability, derived from the adult Affective Lability Scale that was specifically designed for adults with BD. It yields a total score as well as an angry/depressed factor and a disinhibited/impersistent factor. Item scores range from 0 to 4 and higher scores indicate higher affective lability.
Dialectical Behavior Therapy Barriers to Implementation | 12 months to 18 months
  The Dialectical Behavior Therapy Barriers to Implementation (DBT-BTI) is a 26-item self-report survey that assesses barriers to DBT implementation in four domains: team, direction/motivation, theoretical position/philosophy, and administrative/structural problems. It is a yes/no questionnaire and higher scores indicate higher challenges in implementation. To be completed by DBT therapist participants.
Dialectical Behavior Therapy Barriers to Implementation | 18 months to 24 months
  The Dialectical Behavior Therapy Barriers to Implementation (DBT-BTI) is a 26-item self-report survey that assesses barriers to DBT implementation in four domains: team, direction/motivation, theoretical position/philosophy, and administrative/structural problems. It is a yes/no questionnaire and higher scores indicate higher challenges in implementation. To be completed by DBT therapist participants.
Barriers and Facilitators Assessment Instrument (name of scale) | 12 months to 18 months
  Therapists will complete this well-validated and widely used measure, and is the only measure available that is designed to assess barriers and facilitators at each of the levels proposed within one instrument.
Barriers and Facilitators Assessment Instrument (name of scale) | 18 months to 24 months
  Therapists will complete the Barriers and Facilitators Assessment Instrument which is a well-validated and widely used measure, and is the only measure available that is designed to assess barriers and facilitators at each of the levels proposed within one instrument. It is a 16 item Likert scale questionnaire ranging from 1 to 6 with some items being reverse scored. High scores generally indicate challenges to implementation.
Implementation Climate Scale | 12 months to 18 months
  The Implementation Climate Scale will enable the team to document relevant organizational processes the aid in implementation of this treatment and provide a context for other evidence-based treatment dissemination studies. This is a Likert scale from 0 to 4 with low scores indicating challenges with implementation.
Implementation Climate Scale | 18 months to 24 months
  The Implementation Climate Scale will enable the team to document relevant organizational processes the aid in implementation of this treatment and provide a context for other evidence-based treatment dissemination studies. This is a Likert scale from 0 to 4 with low scores indicating challenges with implementation.
Change in therapist self-assessment | Every month for three years through study completion, an average of 36 months.
  The Dialectical Behavior Therapy (DBT) Therapist Self-Assessment will allow for DBT therapists to provide subjective appraisals of their own level of comfort and confidence in applying the treatment. It also assesses the need for additional supervision from the study supervisor, consultant, and/or peer. Scores range from 1 to 7 on a Likert scale and high scores indicate high therapist level of comfort in implementing the treatment.
Number of therapy sessions | At the end of study completion (three years)
  The DBT Therapy Tracking Form will be used to document the date of the therapy session, type of session, session duration, content, and scheduled date for next therapy visit. This form will be completed by the DBT study therapist after each therapy session.
Frequency of therapy sessions | At the end of study completion (three years)
  The DBT Therapy Tracking Form will be used to document the date of the therapy session, type of session, session duration, content, and scheduled date for next therapy visit. This form will be completed by the DBT study therapist after each therapy session.
Type of therapy sessions | At the end of study completion (three years)
  The DBT Therapy Tracking Form will be used to document the date of the therapy session, type of session, session duration, content, and scheduled date for next therapy visit. This form will be completed by the DBT study therapist after each therapy session.
Reasons for continuing or not continuing in treatment | 12 months
  Participants and study therapists will be asked to complete the Dialectical Behavior Therapy Continuation Questionnaire to assess reasons for continuing or not continuing to proceed with the DBT treatment. Items are rated from 1 (strongly disagree) to 7 (strongly agree)
Change in number of hours of supervision | At the end of study completion (three years)
  The Therapist Supervision Hours Log will be completed by the DBT study therapist for all supervision received on study cases. This form includes date of supervision, duration of supervision, and type of supervision.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin I Goldstein, MD, PhD, Principal Investigator — Sunnybrook Research Insitute
Locations (2):
- Canada (2):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Centre for Addiction and Mental Health, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No